CLINICAL TRIAL: NCT07388641
Title: An Innovative Combined Psychosocial Intervention to Improve Productive Community Integration in Homeless-experienced Veterans
Brief Title: Improving Productive Community Integration in Homeless-experienced Veterans
Acronym: MI-CBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRD4-008-25M; 1I01RD000643-01A1 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Homeless Persons
Keywords: motivation; motivational interviewing; psychosocial intervention; work; community integration
MeSH Terms: interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Random assignment to experimental psychosocial treatment of active control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessments will be done by staff members who are entirely unaware of the treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MI-CBT (Experimental): Combination of Motivational Interviewing and Cognitive Behavioral Therapy
  Interventions: Other: Motivational Interviewing and Cognitive Behavioral Therapy
- Health Lifestyles (Active Comparator): An educational program that instructs participants on important concepts in nutrition, exercise, and stress management.
  Interventions: Other: Healthy Behavior Training

INTERVENTIONS:
Other: Motivational Interviewing and Cognitive Behavioral Therapy — Psychosocial intervention to increase motivation for work and productive activities
  Other Names: MI-CBT
  Arms: MI-CBT
Other: Healthy Behavior Training — An educational program on nutrition, exercise, and stress management.
  Other Names: Healthy Lifestyles
  Arms: Health Lifestyles

SUMMARY:
The VA has been focused on reducing the number of homeless Veterans nationally. However, it has been very difficult to increase the level of productive activities--including work, school, and training--for homeless-experienced Veterans (HEVs), even when the VA provides substantial case management and support services in addition to housing. The overarching aim of this proposed treatment project is to validate an innovative psychosocial intervention (a combination of Motivational Interviewing and Cognitive Behavioral Therapy; MI-CBT) that is designed to enhance motivation and increase productive community integration in Veterans who have experienced homelessness. The efficacy of this new intervention will be evaluated in a randomized control trial that includes 24 weeks of active treatment, and a follow up assessment, compared with a control condition. The results of the proposed study will have clinical and functional impact for Veterans by helping HEVs to achieve fuller community integration.

DETAILED DESCRIPTION:
Significance to the VA: The VA has been heavily focused on reducing the number of homeless Veterans nationally. However, it has been very difficult to increase the level of productive activities--including work, school, and training--for homeless-experienced Veterans (HEVs), even when the VA provides substantial case management and support services in addition to housing. The overarching aim of this proposed project is to validate a recovery-oriented psychosocial intervention that is designed to reduce motivational impairments and increase productive community integration in Veterans who have experienced homelessness and are now housed.

Innovation and Impact: The work in two randomized controlled trials (RCT) has shown that an innovative psychosocial intervention, Motivational Interviewing combined with Cognitive Behavioral Therapy (MI-CBT), significantly increases motivation to achieve personally-relevant functional goals compared with a control procedure. However, the investigators do not know whether this new psychosocial intervention can specifically improve productive aspects of community integration which tend to be most resistant to change. Further, the investigators do not understand the mechanisms through which treatments achieve their benefits. The results of the proposed study will have substantial clinical and functional impact for Veterans by helping HEVs to achieve fuller community integration. The findings will also have the potential to influence the types of psychosocial interventions that are being used in Homeless Programs throughout the VA.

Specific Aims: The proposed project has two aims. Aim 1 is to examine the effects of MI-CBT versus a Healthy Lifestyles control intervention on two primary measures (a proximal outcome of motivation and more distal outcome of behavior) related to productive community integration in HEVs over the 24 weeks of active treatment (i.e., 12 weeks of weekly treatment and 12 weeks of monthly boosters). Aim 2 is to examine the treatment effects of MI-CBT versus the control intervention on a secondary outcome measure of effort allocation. The project has Exploratory Aims to assess whether effort allocation is a mediator of observed changes in motivation and productive behavior and to evaluate whether baseline length of housing is a moderator of the treatment effects.

Methodology: The aims will be evaluated in an RCT that includes 24 weeks of active treatment (group sessions weekly for the first half and boosters every 4 weeks thereafter). A follow up assessment will be conducted at 36 weeks to assess durability. The study will include a total of 106 HEVs who are not involved in jobs, school, or training at their baseline assessment. Participants will be randomly assigned 1:1 to MI-CBT or to an active control condition. There will be two primary outcome measures: the proximal treatment target will be motivation for productive activities; the distal target will be community integration based on average hours of productive activity per week. A secondary outcome will be a measure of effort allocation based on performance on an effort-based decision-making task.

Path to Translation / Implementation: In the proposed RCT, HEVs will be randomly assigned to an innovative psychosocial intervention to improve their productive community activities. It is an efficacy study and is considered a T2-A: Phase II trial which is intended to determine the efficacy of therapy in patients. If the proposed project is successful, the subsequent study would be a larger, multi-site RCT in a broader sample of HEVs. That would move the aims into T2-B: Phase III larger clinical trials to establish efficacy and optimal use in humans.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* fluent in English
* history of homelessness and currently housed through VA HUD-VASH housing programs
* expressed willingness to work on a school, work, or training goals

Exclusion Criteria:

* no clinically significant medical, neurological, or physical condition that would interfere with providing informed consent or valid assessments
* no visible sign of intoxication on the laboratory assessment visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-08-03 (Estimated); Primary Completion 2030-08-03 (Estimated); Study Completion 2031-08-03 (Estimated)

PRIMARY OUTCOMES:
Action subscale of the University of Rhode Island Change Assessment Scale | baseline, midpoint at 12 weeks, post-treatment at 24 weeks, and follow-up at 36 weeks
  Measure of attitudes and activities related to motivation for productive activities. The range is 8-40 in which higher scores indicate more willingness to change.
Service Use and Resource Form (SURF) | baseline, midpoint at 12 weeks, post-treatment at 24 weeks, and follow-up at 36 weeks
  average number of hours of productive activities per week for past month

SECONDARY OUTCOMES:
Measure of willingness to exert effort on a cognitive task (Deck choice task) | baseline, midpoint at 12 weeks, post-treatment at 24 weeks, and follow-up at 36 weeks
  measure of effort allocation on a cognitive choice task

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Green, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No